CLINICAL TRIAL: NCT00322400
Title: An Open-label, Dose-finding Study to Evaluate the Safety of AMG 706 in Combination With Paclitaxel or Docetaxel as Treatment for Locally Recurrent or Metastatic Breast Cancer
Brief Title: Phase1b to Evaluate Safety of AMG706 in Combination With Paclitaxel or Docetaxel for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050200
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Locally Recurrent and Metastatic Breast Cancer
Keywords: Clinical trial; AMG 706; Anti-angiogenesis; Locally Recurrent; Metastatic; Breast Cancer; VEGF; Angiogenesis Inhibitor; Oral; Multi-kinase Inhibitor; Anti-tumor; PDGF receptor; Paclitaxel; Docetaxel; Targeted Therapy; Oncology; Amgen; c-Kit
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Docetaxel; Paclitaxel; motesanib diphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- B1 (Experimental): AMG 706 50 mg daily + Docetaxel (100 mg/m2 D1 every 21 days)
  Interventions: Drug: Docetaxel; Drug: AMG 706
- A4 (Experimental): 75 mg AMG 706 daily + Paclitaxel (90 mg/m2 on D1, D8 and D15 every 28 days)
  Interventions: Drug: Paclitaxel; Drug: AMG 706
- A1 (Experimental): AMG 706 50 mg daily + Paclitaxel (90 mg/m2 D1, D8, D15 every 28 days)
  Interventions: Drug: Paclitaxel; Drug: AMG 706
- B4 (Experimental): 75 mg AMG 706 daily + Docetaxel (100 mg/m2, D1 every 21 days)
  Interventions: Drug: Docetaxel; Drug: AMG 706
- B5 (Experimental): MTD of AMG 706 + Docetaxel (75mg/m2 D1 every 21 days)
  Interventions: Drug: Docetaxel; Drug: AMG 706
- B3 (Experimental): 100 mg AMG 706 daily + Docetaxel (100 mg/m2 on D1 every 21 days)
  Interventions: Drug: Docetaxel; Drug: AMG 706
- B2 (Experimental): AMG 706 125 mg daily + Docetaxel (100 mg/m2 D1 every 21 days)
  Interventions: Drug: Docetaxel; Drug: AMG 706
- A2 (Experimental): AMG 706 125 mg daily + paclitaxel 90 mg/m2 D1, D8, D15 every 28 days
  Interventions: Drug: Paclitaxel; Drug: AMG 706
- A3 (Experimental): 100 mg AMG 706 daily + Paclitaxel (90 mg/m2 on D1, D8, and D15 every 28 days)
  Interventions: Drug: Paclitaxel; Drug: AMG 706

INTERVENTIONS:
Drug: Docetaxel — Subjects assigned to Arm B, cohorts will receive 75 or 100 mg/m2 of docetaxel (based on cohort assignment) on Day 1 repeated every 21 days (1 cycle). AMG 706 will be administered concurrently on Days 3-21 of Cycle 1, and Days 1-21 of Cycle 2 and beyond.
  Arms: B1; B2; B3; B4; B5
Drug: Paclitaxel — Subjects assigned to Arm A will receive 90 mg/m2 of paclitaxel on Days 1, 8 and 15 repeated every 28 days (1 cycle). On Arm A, AMG 706 will be concurrently administered on Days 3-28 of Cycle 1, and Days 1-28 of Cycle 2 and beyond.
  Arms: A1; A2; A3; A4
Drug: AMG 706 — Subjects assigned to Arm A will receive AMG 706 at 50, 75, 100 or 125 mg daily (based on cohort assignment) on Days 3-28 of Cycle 1, and Days 1-28 of Cycle 2 and beyond in combination wth paclitaxel 90 mg/m2. Paclitaxel will be administered on Days 1, 8 and 15 every 28 days.
  Subjects assigned to Arm B will receive AMG 706 at 50, 75, 100 or 125 mg daily(based on cohort assignment) on Days 3-21 of Cycle 1, and Days 1-21 of Cycle 2 and beyond in combination with docetaxel. Docetaxel will be administered at either 75 mg/m2 or 100 mg/m2 on Day 1 every 21 days.

SUMMARY:
This open-label, dose-finding, multi-center study is designed to determine the safety and the maximum tolerated dose of AMG 706 given once daily in combination with either weekly paclitaxel (Arm A) or once-every-3 week docetaxel (Arm B) in subjects with locally recurrent or metastatic breast cancer. Secondarily, this study will evaluate the pharmacokinetic (PK) profile of AMG 706 in both treatment arms, the PK profile of paclitaxel in Arm A and the PK profile of docetaxel in Arm B. Additionally, this study will assess objective tumor response and duration of response. Exploratory endpoints include the investigation of potential biomarker development and to assess the effects of genetic variation in drug metabolism genes, cancer genes and drug target genes on subject response to AMG 706 in combination with paclitaxel or docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Female 18 years of age or older.
* Adequate hematologic, renal and hepatic function.
* Competent to comprehend, sign, and date an IRB-approved informed consent form.
* Subjects of childbearing potential and sexually active must provide a negative pregnancy test and use accepted and effective method of contraception.

Exclusion Criteria:

* Prior taxane-containing treatment within 6 months prior to enrollment.
* Prior treatment including chemotherapy and/or endocrine therapy discontinued < 21 days prior to enrollment.
* More than one prior systemic chemotherapy for locally recurrent or metastatic breast cancer.
* Current or prior history of central nervous system metastases.
* History of arterial or venous thrombosis within 1 year prior to enrollment.
* History of bleeding diathesis or bleeding within 14 days prior to enrollment.
* Radiation therapy to a significant portion of bone marrow or prior history of high-dose chemotherapy requiring bone marrow or stem cell support.
* Hypersensitivity to paclitaxel, docetaxel, or drugs using the vehicle cremophor.
* Prior VEGFr targeted therapies within 30 days of enrollment.
* Any anticoagulant therapy within 7 days prior to enrollment, except for warfarin of less than 2mg per day.
* Clinically significant cardiac disease including myocardial infarction or other cardiovascular related event within 1 year before enrollment.
* Uncontrolled hypertension (systolic >150 mmHg; diastolic > 90 mmHg).
* Known HIV positive, hepatitis C positive or hepatitis B surface antigen positive.
* Prior bevacizumab or trastuzumab therapy within 12 weeks of enrollment.
* Non-healing wound, ulcer or fracture.
* Known history of prior episodes of cholecystitis, prior biliary procedure or prior or ongoing biliary disease.
* Unable to take oral medications.
* Not recovered from previous therapies.
* Major surgery within 28 days prior to enrollment.
* Prior malignancy unless treated with curative intent and without evidence of disease for greater than 3 years before enrollment.
* Peripheral neuropathy grade > 1 per CTCAE version 3.0

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-03; Primary Completion 2009-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Cycle 1 of treatment. For Arm A, 1 cycle = 28 days. For Arm B, 1 cycle = 21 days

SECONDARY OUTCOMES:
Pharmacokinetics of AMG 706 when administered with paclitaxel (Arm A) or docetaxel (Arm B) | Cycle 1 (Arms A and B) and Cycle 2 Arm B only)
Pharmacokinetics of paclitaxel (Arm A) when administered with AMG 706 | Cycle 1, D1 and D8 for subjects in Arm A only
Pharmacokinetics of docetaxel (Arm B) when administered with AMG 706 | Cycles 1 and 2 for subjects in Arm B only
Incidence of adverse events and clinical laboratory abnormalities not defined as DLTs | From study entry through 30 days post discontinuation of study treatment
Objective tumor response (complete or partial response) according to modified RECIST | Subjects in Arm A: every 8 weeks until discontuation. Subjects in Arm B:every 6 weeks until discontinuation.
Duration of response (calculated for those subjects who respond): time from first objective tumor response to objective disease progression or death. | Subjects in Arm A: every 8 weeks until discontuation. Subjects in Arm B:every 6 weeks until discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] De Boer RH, Kotasek D, White S, Koczwara B, Mainwaring P, Chan A, Melara R, Ye Y, Adewoye AH, Sikorski R, Kaufman PA. Phase 1b dose-finding study of motesanib with docetaxel or paclitaxel in patients with metastatic breast cancer. Breast Cancer Res Treat. 2012 Aug;135(1):241-52. doi: 10.1007/s10549-012-2135-0. Epub 2012 Jul 29. PMID 22872523
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com